CLINICAL TRIAL: NCT01243489
Title: CRESCENDO (Compliance: Role Emerges for Success in CML: Evaluation aND Optimisation): A Prospective, Multi-center, Phase IV Study to Assess the Compliance in Patients With Philadelphia Chromosome-positive (Ph+) and/or BCR-ABL Positive Chronic Myelogenous Leukaemia (CML) Under Long-term Imatinib Therapy
Brief Title: Compliance: Role Emerges for Success in Chronic Myelogenous Leukaemia (CML): Evaluation aND Optimisation
Acronym: Crescendo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: Crolll Gmbh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSTI571ADE75T; 2010-018339-16 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Chronic Myelogenous Leukemia (CML)
Keywords: CML; compliance; compliance supporting measures; complete cytogenetic response; mayor molecular remission; Philadelphia chromosome; BCR-ABL; Imatinib; tyrosine kinase inhibitor; smart blister
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Patient Compliance; Philadelphia Chromosome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient diary (Other): compliance supporting measure: patients uses patient diary from month 6 to 12
  Interventions: Other: compliance supporting measures
- Information service "Leben mit CML" (Other): compliance supporting measure: patient uses the Information service "Leben mit CML"
  Interventions: Other: compliance supporting measures

INTERVENTIONS:
Other: compliance supporting measures — Patients will be treated for a total of 12 months, 6 months without and 6 months with compliance supporting measures. Patient can choose between an information service "Leben mit CML" or the use of a daily diary

SUMMARY:
This study on patient's compliance in clinical workaday life aims to assess and to improve CML treatment in Germany by means of adherence supporting measures and to increase adherence awareness by physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years) CML patients in the chronic phase
* Medical history of cytogenetically confirmed CML-CP by the presence of the Philadelphia chromosome on bone marrow aspirates (a minimum of 20metaphases is required; FISH cannot be used); Philadelphia chromosome negative but BCR- ABL-positive CML patients can be included
* ECOG performance status of < 2
* Imatinib treatment for at least 1 year and showing CCyR or MMR
* Prior treatment with chemotherapeutics such as hydroxyurea or interferon- alpha is allowed
* Prior periods of accelerated phases are allowed
* Negative pregnancy test for female patients of childbearing potential within 7 days before initiation of study drug
* Ability to understand and willingness to sign a written informed consent document prior to any study related screening procedures
* Written informed consent, including the consent to be called for interviews by the external, neutral institution.

Exclusion Criteria:

* Patients with prior blast crisis or stem cell transplantation
* Patients with severe medical condition(s) that in the discretion of the investigator prohibits participation in the study (e.g., clinically significant heart diseases, uncontrolled diabetes, active or uncontrolled infection, impaired gastrointestinal function/diseases)
* Treatment with drugs or substances, especially those known to modify the cytochrome P450 activity, should be either discontinued or exchanged by different medication (see link for complete list of these medications: http://medicine.iupui.edu/flockhart/table.htm.)
* Pregnant or breastfeeding women
* Male or female of childbearing potential unwilling to use contraceptive precautions throughout the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Patients compliance | 12 months
  To assess patients compliance before and after intervention by comparison of the number of imatinib (Glivec®) tablets taken before and after intervention

SECONDARY OUTCOMES:
Compliance | 12 months
  to correlate the compliance assessed by pill count (conventional pill count and pill count using SmartBlister in selected centers) with the results obtained by the questionnaires and interviews
efficacy of imatinib | 12 months
  to monitor the efficacy of imatinib as assessed by cytogenetics and PCR testing (BCR-ABL load, % IS)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Professor, MD, Principal Investigator — Universitätsklinikum Jena, Klinik für Innere Medizin II
Locations (23):
- Germany (23):
  - Onkologische Schwerpunktpraxis Celle, Celle
  - Onkozentrum Dresden, Gemeinschaftspraxis Dres. Göhler & Dörfel, Dresden
  - Gemeinschaftspraxis Hämatologie - Onkologie, BAG Freiberg-Richter / Jacobasch / Illmer / Wolf, Dresden
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Erfurt
  - St.-Antonius-Hospital, Klinik für Hämatologie und Onkologie, Eschweiler
  - IFS - Interdisziplinäres Facharztzentrum Sachsenhausen, Frankfurt
  - Hämato-Onkologische Schwerpunktpraxis, Dres. Michael Metz, Andreas Ammon, Dirk Meyer, Göttingen
  - MediProjekt, Gesellschaft für Medizinstatistik und Projektentwicklung, Hanover
  - Praxis für Innere Medizin, Onkologie und Hämatologie, Dr. Hahnfeld, Jena
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena
  - Gemeinschaftspraxis Dr. Siehl, Dr. Söling und Prof. Dr. Hirschmann, Kassel
  - Gemeinschaftspraxis, Dres. Neise, Lollert, Krefeld
  - Gemeinschaftspraxis, Dres. Ursula Vehling-Kaiser, Doris Greif, Landshut
  - Internistische Schwerpunktpraxis Dr. Tschechne, Lehrte
  - Onkologische Schwerpunktpraxis, Dres. Uthgenannt, Kisro, Weber, Lübeck
  - Onkonet GbR, Praxis Dres. Weidenbach & Balser, Marburg
  - Hämatologisch onkologische Schwerpunktpraxis, Mayen
  - Nordbadpraxis, München
  - Hämato - Onkologische Praxisgemeinschaft, Dr. Schmidt, München
  - Praxis Dr. Walter, Paderborn
  - Fachärzte für Innere Medizin, Hämatologie & Onkologie Rostock, Rostock
  - Hämatologisch-Onkologische Gemeinschaftspraxis Würselen, Würselen
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie und Internistische Onkologie, Würzburg